CLINICAL TRIAL: NCT06383039
Title: The Effect of Transcranial Direct Current Stimulation on Balance on Supplementary Motor Area and Cerebellum in Healthy Individuals
Brief Title: Transcranial Direct Current Stimulation and Balance
Acronym: tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Soy (Other)
Responsible Party: Sponsor-Investigator, Zeynep Soy, Principal Investigator, Medipol University
Organization: Medipol University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ZSoy
Record Dates: First submitted 2024-02-02; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Balance
Keywords: tDCS; balance; supplementary motor area; cerebellum
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: All participants received 3 different interventions at different times.
Who Masked: Participant
Masking Description: Participants were not informed which type of current was applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sham tDCS (Sham Comparator): Sham transcranial Direct Current Stimulation
  Interventions: Device: Transcranial Direct Current Stimulation
- sma tDCS (Active Comparator): Anodal-supplementary motor area transcranial Direct Current Stimulation
  Interventions: Device: Transcranial Direct Current Stimulation
- cerebellar tDCS (Active Comparator): Anodal-cerebellar transcranial Direct Current Stimulation
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Evaluations will be made in the presence of a physiotherapist. Individuals; For demographic information
  • Demographic Information Form
  For Static Balance Evaluation:
  * Wii-Fit
  * Balance Error Scoring System
  For Dynamic Balance Assessment:
  * Star Balance Test
  * Timed Get Up and Go Test

SUMMARY:
Postural control is an adaptive sensorimotor process involving continuous integration of sensory information from three channels. These; visual, somatosensory (proprioceptive) and vestibular senses. The study will be carried out at Istanbul Medipol University. 30 healthy individuals between the ages of 18-25 will be included. To each individual Anodal-supplementary motor area tDCS, Anodal-cerebellar tDCS, Sham tDCS applications will be cross-applied. tDCS application will take 20 minutes and each individual will receive 3 sessions in total. There will be a 72-hour rest period between sessions. Individuals assessed with Demographic Information Form for demographic information, Wii-Fit and Balance Error Scoring System for Static Balance Evaluation, Star Balance Test and Timed Get Up and Go Test for Dynamic Balance Assessment. The aim of this study is to investigate the effect of transcranial direct current stimulation applied on the supplementary motor area and cerebellum on static and dynamic balance in healthy individuals.

DETAILED DESCRIPTION:
Postural control is an adaptive sensorimotor process involving continuous integration of sensory information from three channels. These; visual, somatosensory (proprioceptive) and vestibular senses. The cerebellum plays an important role in the planning, initiation and stability of movements, as well as in postural control and balance. The Supplementary Motor Area (SMA) is a section of the cortex that plays a major role in planning both simple and complex motor movements; It has many functions such as sequence of movements (turning one's hand before picking up an object), learning (learning a new balance task), acquiring grammar. The SMA is somatotopic organized and has direct reciprocal connections with the primary motor cortex (M1). Independent of the primary motor cortex (M1), the SMA is thought to play a crucial role in planning motor actions before movement begins. It also contributes to the planning of all body movements together with the basal ganglia and cerebellum during challenging balance tasks.

Modulation of neural regions underlying balance control may be a potential alternative for therapy. Transcranial direct current stimulation (tDCS) is a non-invasive and safe tool that can modulate cerebellar activity. tDCS is an easy, inexpensive and portable device to implement. There are 3 different types of stimulation. While anodal stimulation promotes neural excitability by causing subthreshold depolarization, cathodal stimulation inhibits neural activity, and in addition, anode-cathode application, in which two types of stimulation are used together, provides both facilitation and inhibition according to electrode placement. In a study conducted by Foerster et al. in healthy individuals in 2017, it was found that cerebellar tDCS increased balance stability, and in a study by Ehsani et al. in healthy individuals over 60 years of age in 2017, cerebellar tDCS increased the Berg Balance balance score. In a study conducted by Steiner et al. in 2016 in which cerebellar tDCS was applied to young individuals, it was observed that the trunk deviation angle during balance was decreased in men, while a similar study by Inukai et al. showed a decrease in oscillation after cathodal cerebellar tDCS.

There are studies showing that tDCS applied to the supplementary motor area has positive contributions to balance. It has been shown by Nomura et al. that tDCS applied to the supplementary motor area in healthy individuals causes a significant increase in balance.

There is no study comparing supplementary motor area and cerebellar area application in healthy individuals where tDCS is applied.

In line with these studies, the aim of this study is:

To investigate the effect of transcranial direct current stimulation applied on the supplementary motor area and cerebellum on static and dynamic balance in healthy individuals.

The study will be carried out at Istanbul Medipol University. 30 healthy individuals between the ages of 18-25 will be included.

To each individual:

1. Anodal-supplementary motor area tDCS
2. Anodal-cerebellar tDCS
3. Sham tDCS applications will be cross-applied. tDCS application will take 20 minutes and each individual will receive 3 sessions in total. There will be a 72-hour rest period between sessions. Evaluations will be made at the beginning and will be repeated immediately after tDCS applications.

Inclusion Criteria:

* No neurological, sensory, motor, visual or cognitive impairment,
* Volunteering to participate in the study,
* Being between the ages of 18-25,
* To have formal education at the university.

Exclusion Criteria:

• Being diagnosed with a psychological disorder.

Evaluations will be made in the presence of a physiotherapist. Individuals; For demographic information

• Demographic Information Form

For Static Balance Evaluation:

* Wii-Fit
* Balance Error Scoring System

For Dynamic Balance Assessment:

* Star Balance Test
* Timed Get Up and Go Test

It will be evaluated with IBM SPSS "Statistical Package for Social Sciences".

ELIGIBILITY:
Inclusion Criteria:

* No neurological, sensory, motor, visual or cognitive impairment,
* Volunteering to participate in the study,
* Being between the ages of 18-25,
* To have formal education at the university.

Exclusion Criteria:

* Being diagnosed with a psychological disorder.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2023-05-13 (Actual)

PRIMARY OUTCOMES:
Demographic Information Form | 4 months
  Demographic Information Form includes the patient's personal information, sociodemographic and physical characteristics.İt includes: name, surname, date of the birth, using cigarette / alcohol, presence presence of disease, using drugs
Wii-Fit | 4 months
  Nintendo Wii Fit Balance Evaluation was carried out in a darkened room with no light. In this setup, the Nintendo Wii Fit image was projected on the wall with a projector. The patient's birth year and height were recorded according to the device's instructions. The patient's weight was calculated in centimeter by the device. The patient was taught how to step on the board. First, the patient was asked to stand looking straight ahead without moving, and the center of gravity on the right and left foot was calculated as a percentage. Then the patient's body mass index was calculated in kg/m^2. Afterwards, the patient was asked to step in the middle of the balance board with one foot and maintain this position for 30 seconds. A single-leg stabilization test was performed separately for both feet and the results were recorded as a percentage.
balance error scoring system | 4 months
  2 different surfaces and 3 stance positions . Normal floor is used for flat surface, foam block is used for foam surface. Subjects apply the 6 conditions of the test in the following order: flat surface with two legs support, one foot support and tandem stance position; sponge surface with two legs support, one foot support and tandem stance. The duration of each position was measured by a smart watch for approximately 20 seconds. Each mistake made by individuals within 20 seconds was recorded as 1 point. Six different situations counted as errors are as follows: - Pulling the arms over the iliac crest - Opening the eyes - Taking a step, stumbling or falling - Flexing or abducting the hip joint more than 30° - Lifting the foot or heel off the ground - More than five seconds out of the test position staying too long. Error scores were calculated separately for each position and the total error score was obtained by adding the scores. Higher score indicates worse balance
star excursion balance test | 4 months
  On the determined floor, 4 strips cut in 2 meters length are adhered to form 45 degree angles between them. The participant waits in the middle of the star shape (the point where the lines intersect).The participant reaches as far as she can reach with her foot.Then the other line is passed and a total of 8 lines are completed in this way.At the end of each distance, a mark was made with a pencil so that you could measure it later. Highest score was obtained from 3 reaches in each direction.
Time Up & Go Test | 4 months
  3 meters area is determined in front of the chair. The patient is asked to get up from his seat and go to the designated place and sit down again. The time is recorded in seconds. shorter time indicates better balance

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elsner B, Kwakkel G, Kugler J, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving capacity in activities and arm function after stroke: a network meta-analysis of randomised controlled trials. J Neuroeng Rehabil. 2017 Sep 13;14(1):95. doi: 10.1186/s12984-017-0301-7. PMID 28903772
- [Background] Hayduk-Costa G, Drummond NM, Carlsen AN. Anodal tDCS over SMA decreases the probability of withholding an anticipated action. Behav Brain Res. 2013 Nov 15;257:208-14. doi: 10.1016/j.bbr.2013.09.030. Epub 2013 Sep 21. PMID 24064279
- [Background] Peterka RJ. Sensorimotor integration in human postural control. J Neurophysiol. 2002 Sep;88(3):1097-118. doi: 10.1152/jn.2002.88.3.1097. PMID 12205132
- [Background] Hupfeld KE, Ketcham CJ, Schneider HD. Transcranial direct current stimulation (tDCS) to the supplementary motor area (SMA) influences performance on motor tasks. Exp Brain Res. 2017 Mar;235(3):851-859. doi: 10.1007/s00221-016-4848-5. Epub 2016 Dec 1. PMID 27909747